CLINICAL TRIAL: NCT00895570
Title: Sleep Restriction, Impaired Glucose Metabolism, and Performance: The Effects of Modafinil to Counteract the Adverse Metabolic Consequences of Sleep Restriction
Brief Title: The Effects of Modafinil to Counteract the Adverse Metabolic Consequences of Sleep Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Dr. Orfeu Buxton, Ph.D., Brigham & Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C1538/6032/ES/US
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Sleep Restriction; Impaired Glucose Metabolism
Keywords: sleep restriction; glucose metabolism; modafinil; euglycemic clamp; insulin sensitivity; insulin release
MeSH Terms: conditions — Insulin Resistance | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modafinil (Experimental): During each day of the 7-day sleep restriction phase of the study modafinil was administered (200 mg tablet at 0600, and a second dose of 100 mg tablet at 1300).
  Interventions: Drug: modafinil
- Placebo (Placebo Comparator): During each day of the 7-day sleep restriction phase of the study a sugar pill was administered.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: modafinil — During each day of the 7-day sleep restriction phase of the study modafinil was administered (200 mg tablet at 0600, and a second dose of 100 mg tablet at 1300).
  Other Names: Provigil
  Arms: Modafinil
Drug: placebo — During each day of the 7-day sleep restriction phase of the study a sugar pill was administered.
  Arms: Placebo

SUMMARY:
The purpose of the study is to examine the effects of sleep and modafinil on how the body processes glucose.

DETAILED DESCRIPTION:
The occurrence and diagnosis of DM2 and its complications is increasing, leading to rising treatment costs that represent a considerable portion of the U.S. health care budget. Although treatment of impaired glucose tolerance (IGT) is not common, an IGT diagnosis increases the likelihood of progression to DM2. Careful attention to glycemic control is a primary treatment goal for DM2 patients, as glucose control reduces the severity of microvascular, macrovascular, and other complications.

Recent research has indicated that sleep loss could be a previously unrecognized risk factor for DM2. As sleep restriction has become an endemic condition in developed countries, it is possible that sleep loss contributes to the recent epidemic of DM2. Protecting sleep by increasing sleep duration and quality in DM2 and IGT patients may provide an inexpensive, relatively easy to implement intervention to reduce the risk of disease onset or delay disease progression by improving glucose tolerance. Furthermore, measurement of endocrine, metabolic, and cardiovascular parameters in the proposed studies may provide insights into the mechanisms by which sleep extension improves glucose tolerance under pathophysiological conditions.

The proposed study examines and quantifies in adults the link between insufficient sleep and increased insulin resistance, impaired insulin secretion, and reduced non-insulin-dependent glucose utilization by the sleepy brain. The proposed study capitalizes upon the unique pharmacological characteristics of modafinil to reverse excessive sleepiness to address the mechanisms by which sleep restriction may impact metabolism via excessive sleepiness. This study may lead to countermeasures to the adverse health impact of chronic insufficient sleep, an increasingly common lifestyle that may ultimately contribute to the development of the Metabolic Syndrome or DM2 via alterations of glucose metabolism and brain glucose utilization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have also demonstrated a full understanding of the requirements and demands of the study.
* Individuals must have been willing to follow a regular sleep-wake schedule.

Exclusion Criteria:

* Sleep/wake history. During completion of the preliminary telephone and written screening questionnaires, potential volunteers were asked a number of questions about their present, past and desired habitual sleep/wake schedule, including their habitual and desired bedtimes, wake-times, and nap times. Those potential volunteers with a history of night-work in the preceding 3-year period or travel across >2 time zones in the 3 months prior to the study were excluded.
* Individuals who are unable or unwilling to follow a regular sleep-wake schedule were excluded from the study.
* Drug/Alcohol Use. Volunteers must have been drug-free (including nicotine) and with moderate or no use of caffeine or alcohol for the entire duration of the study. No medications (prescription or over the counter) that significantly affect circadian rhythms, endocrine physiology, or sleep were allowed. They must have had no history of drug or alcohol dependency. No caffeine or alcohol were allowed for one week prior to or during the inpatient portion of the protocol. A comprehensive toxicological analysis of blood and urine for prescription medication, non-prescription medication, drugs of abuse, and caffeine, nicotine and alcohol metabolites was carried out for verification of reported non-use during the initial screening and on the day of admission to the laboratory for verification.
* Evaluation of Medical Suitability. Only healthy, non-obese men were selected for this study. Subjects must have been free from any acute, chronic or debilitating medical conditions. Normality was established on the basis of clinical history, electrocardiogram, clinical biochemical screening tests of blood and urine, and a physical examination conducted by a licensed physician. Any subject with symptoms of active illness (e.g., fever, leukocytosis, hypertension) was excluded from study. Given the wide range of illnesses that are encountered in medical practice, it would not be possible to provide a comprehensive list of each and every disease that could serve as grounds for exclusion for the subject. However, the following is a list of illnesses that would certainly have been grounds for exclusion: Chronobiologic Disorders, Sleep Disorders, Diseases of the Cardiovascular System, Disorders of the Kidney and Urinary Tract, Infectious Diseases, Disorders of the Gastrointestinal System, Disorders of the Immune System, Connective Tissue and Joints, Disorders of the Hematopoietic System, Neoplastic Diseases, Endocrine and Metabolic Diseases, Neurologic Disorders; significant impairments of the visual system.
* Evaluation of Psychiatric/Psychological Suitability. Each potential volunteer completed a series of psychological questionnaires received a comprehensive psychological examination by a clinical psychologist experienced with the psychological screening for the subjects in our studies. Individuals with evidence of psychopathology on standardized questionnaires or in a structured interview were excluded from study. Individuals with a history of psychiatric illnesses or psychiatric disorders were excluded. Individuals who are unaware of specific psychiatric diagnoses who have a history of having been treated with antidepressant, neuroleptic medications or major tranquilizers were excluded from study. However, a personal history of limited prior counseling or psychotherapy (e.g., for adjustment reactions) was not necessarily exclusionary. Potential subjects were evaluated for Axis II personality types that might interfere with protocol compliance or with their personal ability to tolerate the conditions of the study, such as temporal isolation and confinement.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity measured with euglycemic hyperinsulinemic clamp | Following 3 nights of a continued 'sleep replete' period with 10 hours/night of time in bed and again following 7 days sleep restricted to 5 hrs time in bed/night

SECONDARY OUTCOMES:
Insulin release (i.e., pancreatic beta cell function) measured on IVGTT | Following 3 nights of a continued 'sleep replete' period with 10 hours/night of time in bed and again following 7 days sleep restricted to 5 hrs time in bed/night
Glucose effectiveness measured using an IVGTT, clamp | Following 3 nights of a continued 'sleep replete' period with 10 hours/night of time in bed and again following 7 days sleep restricted to 5 hrs time in bed/night
Biomarkers of Sleep Loss (HbA1c, fructosamine, insulin, glucose, cortisol thyrotropic axis function, lipid metabolism, leptin, ghrelin and cytokine signaling) | Following 3 nights of a continued 'sleep replete' period with 10 hours/night of time in bed and again following 7 days sleep restricted to 5 hrs time in bed/night
Subjective measures of sleepiness and alertness | Every 3 hours while awake during the 12-day inpatient stay
RMR assessed by indirect calorimetry | On the morning and late afternoon of day 4 and 11
Urinary catecholamines levels | Over 24 hours on days 3, 4, 10, 11
Salivary free cortisol | Every 30 minutes in the afternoon of days 3, 4, 10, 11
Neurobehavioral performance | approx very 3 hours during wake in the 12-day inpatient stay

CONTACTS AND LOCATIONS:
Overall Officials: Orfeu M Buxton, Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Buxton OM, Pavlova M, Reid EW, Wang W, Simonson DC, Adler GK. Sleep restriction for 1 week reduces insulin sensitivity in healthy men. Diabetes. 2010 Sep;59(9):2126-33. doi: 10.2337/db09-0699. Epub 2010 Jun 28. PMID 20585000